CLINICAL TRIAL: NCT02563496
Title: An Open Label, Non-comparative, Multicenter Study to Assess the Pharmacokinetics, Safety and Efficacy of Tafenoquine (SB-252263, WR238605) in the Treatment of Pediatric Subjects With Plasmodium Vivax Malaria
Brief Title: A Pharmacokinetics, Safety and Efficacy Study of Tafenoquine (TQ) in Pediatric Subjects With Plasmodium Vivax (P. Vivax) Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113577
Record Dates: First submitted 2015-09-10; First posted 2015-09-30 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Malaria, Vivax
Keywords: pharmacokinetic; pediatric; Tafenoquine; Plasmodium vivax Malaria; G6PD deficiency
MeSH Terms: conditions — Malaria, Vivax; Glucosephosphate Dehydrogenase Deficiency | interventions — tafenoquine; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Tafenoquine 50 mg (Experimental): Subjects with weight band of >=5 to <=10 kilogram (kg) will receive 50 mg tafenoquine on Day 1. Subject may receive CQ per local/national guidelines.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine
- Tafenoquine 100 mg (Experimental): Subjects with weight band of >10 to <=20 kg will receive 100 mg tafenoquine on Day 1. Subject may receive CQ per local/national guidelines.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine
- Tafenoquine 150 mg (Experimental): Subjects with weight band of >10 to <=20 kg will receive 150 mg tafenoquine on Day 1. Subject may receive CQ per local/national guidelines.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine
- Tafenoquine 200 mg (Experimental): Subjects with weight band of >20 to <=35 kg will receive 200 mg tafenoquine on Day 1. Subject may receive CQ per local/national guidelines.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine
- Tafenoquine 300 mg (Experimental): Subjects with weight band of >35 kg will receive 300 mg tafenoquine on Day 1. Subject may receive CQ per local/national guidelines.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine tablet is supplied as film-coated tablet (100 mg, 150 mg, 200 mg and 300 mg) and fast-dispersing film coated tablet (50 mg).
Drug: Chloroquine — Subjects may receive chloroquine according to local/national treatment guidelines.

SUMMARY:
This is a prospective, open-label, multicenter, non-comparative, single arm study of pediatric subjects with Plasmodium vivax (P. vivax) malaria, aged 6 months to <16 years of age. A total of 60 subjects will be enrolled. Potential subjects who are slide-positive for P. vivax will be started by the site on chloroquine (CQ) per local/national guidelines. Sites will have up to 48 hours to obtain consent. Once full consent is provided, all subjects will be screened and, if eligible, receive Tafenoquine (TQ), given as a single dose on Day 1. All study medication should be taken with food. After the treatment period, subjects will attend up to 7 follow-up visits through Day 120 (Days 3, 8, 15, 29, 60, 90 and 120). The main cohort will consist of subjects aged >=2 years to <16 years with no restriction on gender. Subjects will be dosed according to four weight bands. Within the total of 60 enrolled pediatric subjects, a second cohort of up to 6 infants aged >=6 months to <2 years (weighing >=5 kilogram [kg]) will be recruited following completion of a planned first interim analysis. An interim analysis will be conducted once sufficient data from 16 subjects is available to assess pharmacokinetic (PK) and safety parameters. If needed, a second interim analysis will be conducted after a total of 32 subjects have enrolled. The primary objective of this PK bridging study is to adequately characterize the systemic TQ exposure in the pediatric population in order to identify appropriate doses that achieve a similar exposure to that of the TQ adult dose of 300 milligram (mg).

ELIGIBILITY:
Inclusion Criteria:

* Subject is >=2 years to <16 years of age at the time of signing of the assent and/or informed consent. An additional cohort of subjects aged >=6 months to <2 years may be recruited following the first interim analysis.
* The subject has a positive malarial smear for P. vivax.
* The subject has a history of fever within 48 hours prior to enrollment.
* The subject has a glucose 6-phosphate dehydrogenase (G6PD) value (measured by a quantitative spectrophotometric phenotype assay) >=70% of the site median value for G6PD normal adult males.
* The subject has a screening Hb value >=8 gram per decilitre (g/dL).
* The subject has a body weight >=5 kg.
* Males and females are eligible to enter the study. A female is eligible to enter and participate in this study if she is non-pregnant, non-lactating and if she is of: Non-childbearing potential (i.e., premenstrual); or Child-bearing potential, has a negative pregnancy test at screening, and agrees to comply with one of the following during the treatment stage of the study and for a period of 90 days after stopping study medication: Complete abstinence from intercourse for 2 weeks prior to administration of study medication, throughout the study and for a period of 90 days after stopping study medication; Use of combined oral contraceptive consisting of spermicide with either condom or diaphragm; Use of intrauterine device with a documented failure rate of <1% per year; Use of depo provera injection; Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female.
* The subject and/or the subject's parent(s)/legal guardian(s) agree to G6PD genotyping in the context of a subsequent hemolytic anemia AE.
* The subject and parent(s)/legal guardian(s) are willing and able to comply with the study protocol.
* In accordance with regional/local laws and regulations, the parent(s)/legal guardian(s) has given written informed, dated consent; and the subject has given written assent, if applicable, to participate in the study.

Exclusion Criteria:

* The subject has a mixed malaria infection (identified by a malarial smear or rapid diagnostic test).
* The subject has a condition that may affect absorption of study medication, such as severe vomiting (no food or inability to take food during the previous 8 hours).
* The subject has a liver alanine aminotransferase (ALT) >2 time the upper limit of normal (ULN).
* The subject has a clinically significant concurrent illness (for example; pneumonia, meningitis, septicaemia, coagulopathy, severe hemorrhage), pre-existing condition (e.g., renal disease, malignancy, malnutrition, known pre-existing human immunodeficiency virus [HIV]), febrile convulsions prior to consent, or clinical signs and symptoms of severe cardiovascular disease (for example; congenital heart disease).
* The subject has a history of porphyria, psoriasis, or epilepsy.
* The subject has taken anti-malarials (for example; artemisinin-based combination therapies, mefloquine, primaquine, or any other 4- or 8-aminoquinoline) or drugs with antimalarial activity within 30 days prior to study entry.
* The subject has received treatment with any investigational drug within 30 days of study entry, or within 5 half-lives, whichever is longer.
* The subject has taken or will likely require during the study the use of: histamine-2 blockers, antacids, anti-diabetic drugs of the biguanide class (i.e., phenformin, buformin), anti-arrhythmic agents dofetilide, procainamide, pilsicainide.
* The subject has a serum creatinine above the ULN and is currently taking metformin.
* The subject has a history of allergy or intolerance to chloroquine, mefloquine, tafenoquine, primaquine, or to any other 4- or 8-aminoquinoline.
* The subject has previously enrolled in this study.
* The subject has severe P. vivax malaria as defined by world health organization (WHO) criteria

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Montería, Colombia
- Vietnam (2):
  - GSK Investigational Site, Hanoi
  - GSK Investigational Site, Ho Chi Minh City

REFERENCES:
- [Derived] Velez ID, Hien TT, Green JA, Martin A, Sharma H, Rousell VM, Breton JJ, Ernest TB, Rolfe K, Taylor M, Mohamed K, Jones SW, Chau NH, Hoa NT, Duparc S, Tan LK, Goyal N. Tafenoquine exposure assessment, safety, and relapse prevention efficacy in children with Plasmodium vivax malaria: open-label, single-arm, non-comparative, multicentre, pharmacokinetic bridging, phase 2 trial. Lancet Child Adolesc Health. 2022 Feb;6(2):86-95. doi: 10.1016/S2352-4642(21)00328-X. Epub 2021 Dec 3. PMID 34871570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, Phase 2, multicenter study to assess the pharmacokinetics, safety and efficacy of tafenoquine in participants with Plasmodium Vivax Malaria.
Pre-assignment Details: A total of 66 participants were screened, of which 6 participants failed screening. Hence, 60 participants were enrolled in this study. The cohort Tafenoquine 50mg was initiated, but study sites were unable to find any participants who met the inclusion/exclusion criteria for this cohort. Hence, no participants were enrolled in this cohort.
Groups:
- Tafenoquine 50 mg: Participants with weight band of >=5 to <=10 kilogram (kg) were planned to receive 50 milligram (mg) tafenoquine on Day 1. Participants were planned to receive Chloroquine according to local/national guidelines to treat the blood stage of Plasmodium vivax.
- Tafenoquine 100 mg: Participants with weight band of >10 to <=20 kg received 100 mg tafenoquine on Day 1. Participants received Chloroquine according to local/national guidelines to treat the blood stage of Plasmodium vivax.
- Tafenoquine 150 mg: Participants with weight band of >10 to <=20 kg received 150 mg tafenoquine on Day 1. Participants received Chloroquine according to local/national guidelines to treat the blood stage of Plasmodium vivax.
- Tafenoquine 200 mg: Participants with weight band of >20 to <=35 kg received 200 mg tafenoquine on Day 1. Participants received Chloroquine according to local/national guidelines to treat the blood stage of Plasmodium vivax.
- Tafenoquine 300 mg: Participants with weight band of >35 kg received 300 mg tafenoquine on Day 1. Participants received Chloroquine according to local/national guidelines to treat the blood stage of Plasmodium vivax.
Period: Overall Study
Arm/Group | Tafenoquine 50 mg | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
Started | 0 (No participants were enrolled since they didn't meet inclusion/exclusion criteria.) | 14 | 5 | 22 | 19
Completed | 0 | 14 | 5 | 22 | 19
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The tafenoquine 50 mg cohort was initiated, but study sites were unable to find any participants who met the inclusion/exclusion criteria for this cohort. Hence, no participants were enrolled in this cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafenoquine 50 mg | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg | Total
Number analyzed (Participants) | 0 | 14 | 5 | 22 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety Population consisted of all participants who received at least one dose of study medication (tafenoquine).
  Years |  | 4.6 (1.99) | 4.8 (2.05) | 10.2 (1.82) | 12.8 (1.62) | 9.3 (3.80)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population consisted of all participants who received at least one dose of study medication (tafenoquine).
  Participants
    Female |  | 6 | 3 | 8 | 7 | 24
    Male |  | 8 | 2 | 14 | 12 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Safety Population consisted of all participants who received at least one dose of study medication (tafenoquine).
  Participants
    American Indian or Alaskan Native |  | 9 | 0 | 11 | 8 | 28
    Asian: South East Asian Heritage |  | 5 | 5 | 11 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 Extrapolated to Infinite Time (AUC[0-infinity]) of Tafenoquine by Weight Band in Participants Aged >=2 Years to <16 Years (Weighing >=5 kg)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of tafenoquine. Pharmacokinetic parameters were determined using standard non-compartmental methods. AUC(0-infinity) of tafenoquine was evaluated for participants aged >=2 years to <16 years (weighing >=5 kg). Pharmacokinetic (PK) population consisted of all participants with at least one PK sample taken at Days 3, 15, 29 and 60, with accurate dosing and sample time histories.
Time Frame: Days 3, 15, 29 and 60 post dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours*microgram per milliliter
Arm/Group | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
Number analyzed (Participants) | 14 | 4 | 22 | 18
Hours*microgram per milliliter | 85.1 [47.1 to 116.2] | 154.7 [107.4 to 247.1] | 111.4 [73.8 to 143.0] | 120.8 [36.1 to 181.2]

2. Secondary Outcome: Number of Participants With Gastrointestinal Adverse Events
Description: Number of participants experiencing gastrointestinal adverse events including vomiting, abdominal pain, diarrhea, gastrointestinal disorder, epigastric discomfort and nausea were assessed. Number of participants with gastrointestinal adverse events for each treatment group have been presented. Safety Population consisted of all participants who received at least one dose of study medication (tafenoquine).
Time Frame: Up to Day 120
Population: Safety Population. Data is not presented for the cohort Tafenoquine 50 mg; as no participants were enrolled in this cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
Number analyzed (Participants) | 14 | 5 | 22 | 19
Participants
  Vomiting | 2 | 3 | 1 | 6
  Abdominal pain | 0 | 0 | 3 | 0
  Diarrhea | 2 | 0 | 1 | 0
  Gastrointestinal disorder | 0 | 1 | 1 | 0
  Epigastric discomfort | 0 | 0 | 0 | 1
  Nausea | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Hemoglobin Decline From Baseline Over First 10 Days
Description: Glucose-6-phosphate dehydrogenase (G6PD) deficiency is known to be a risk factor for hemolysis in participants treated with 8-aminoquinolines. Blood samples were collected for the evaluation of hemoglobin levels. Hemoglobin decrease of >=30 percent (%) of >30 grams per liter (g/L) from Baseline; or, an overall drop in hemoglobin below 60.0 g/L in the first 15 days of the study were considered as protocol defined serious adverse events (SAEs). Number of participants with hemoglobin decline from Baseline over first 10 days have been presented. Baseline was defined as the latest pre-tafenoquine dose assessment on Day 1.
Time Frame: Baseline and up to Day 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
Number analyzed (Participants) | 14 | 5 | 22 | 19
Participants
  <=20 g/L | 14 | 5 | 21 | 19
  >20 g/L to <=30 g/L | 0 | 0 | 1 | 0
  >30 g/L or >=30% | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/ birth defect, other situations and is associated with liver injury.
Time Frame: Up to Day 120
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
Number analyzed (Participants) | 14 | 5 | 22 | 19
Participants
  Non-SAEs | 10 | 4 | 10 | 13
  SAEs | 0 | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With Worst Case Hematology Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of eosinophils, lymphocytes, platelets and reticulocytes. PCI ranges were >1.5*10^9 (high) cells per liter (cells/L) for eosinophils, <0.5*10^9 cells/L (low) or >4*10^9 cells/L (high) for lymphocytes, <50*10^9 cells/L (low) for platelet count and >1*upper limit of normal (ULN) 10^12 cells/L (high) for reticulocyte count. Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in "To within Range or No Change" category. Participants were counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Baseline value is the latest pre-tafenoquine dose assessment on Day 1.
Time Frame: Baseline (Day 1) and up to Day 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
Number analyzed (Participants) | 14 | 5 | 22 | 19
Participants
  Eosinophils: To Low | 0 | 0 | 0 | 0
  Eosinophils: To within Range or No Change | 12 | 4 | 20 | 18
  Eosinophils: To High | 2 | 1 | 2 | 1
  Lymphocytes: To Low | 0 | 0 | 0 | 0
  Lymphocytes: To within Range or No Change | 9 | 3 | 20 | 16
  Lymphocytes: To High | 5 | 2 | 2 | 3
  Platelet count: To Low | 0 | 0 | 0 | 0
  Platelet count: To within Range or No Change | 14 | 5 | 22 | 19
  Platelet count: To High | 0 | 0 | 0 | 0
  Reticulocyte count: To Low | 0 | 0 | 0 | 0
  Reticulocyte count: To within Range or No Change | 13 | 5 | 18 | 15
  Reticulocyte count: To High | 1 | 0 | 4 | 4

6. Secondary Outcome: Number of Participants With Worst Case Clinical Chemistry Results Relative to PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of clinical chemistry parameters. PCI ranges were >3*ULN international units per liter (IU/L) (alanine aminotransferase [ALT]), >2.5*ULN IU/L (alkaline phosphatase), >3*ULN IU/L (aspartate aminotransferase [AST]), >1.5*ULN micromoles/L (mcmol/L) (bilirubin), >5*ULN IU/L (creatine kinase [CK]), 3*ULN mcmol/L (creatinine), >1.5*ULN mcmol/L (indirect bilirubin), and >11.067 millimoles/L (urea). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "To within Range or No Change" category. Participants were counted twice if participant has values that changed "To Low and To High", so the percentages may not add to 100%. Baseline value is the latest pre-Tafenoquine dose assessment on Day 1.
Time Frame: Baseline (Day 1) and up to Day 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
Number analyzed (Participants) | 14 | 5 | 22 | 19
Participants
  ALT: To Low | 0 | 0 | 0 | 0
  ALT: To within Range or No Change | 14 | 5 | 22 | 19
  ALT: To High | 0 | 0 | 0 | 0
  Alkaline phosphatase: To Low | 0 | 0 | 0 | 0
  Alkaline phosphatase: To within Range or No Change | 14 | 5 | 21 | 19
  Alkaline phosphatase: To High | 0 | 0 | 1 | 0
  AST: To Low | 0 | 0 | 0 | 0
  AST: To within Range or No Change | 14 | 5 | 22 | 19
  AST: To High | 0 | 0 | 0 | 0
  Bilirubin: To Low | 0 | 0 | 0 | 0
  Bilirubin: To within Range or No Change | 14 | 5 | 22 | 19
  Bilirubin: To High | 0 | 0 | 0 | 0
  CK: To Low | 0 | 0 | 0 | 0
  CK: To within Range or No Change | 14 | 5 | 22 | 19
  CK: To High | 0 | 0 | 0 | 0
  Creatinine: To Low | 0 | 0 | 0 | 0
  Creatinine: To within Range or No Change | 14 | 5 | 22 | 19
  Creatinine: To High | 0 | 0 | 0 | 0
  Indirect bilirubin: To Low | 0 | 0 | 0 | 0
  Indirect bilirubin: To within Range or No Change | 14 | 5 | 22 | 19
  Indirect bilirubin: To High | 0 | 0 | 0 | 0
  Urea: To Low | 0 | 0 | 0 | 0
  Urea: To within Range or No Change | 14 | 5 | 22 | 19
  Urea: To High | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Relapse-Free Efficacy at 4 Months
Description: Relapse is defined as positive blood smear with or without vivax malaria symptoms. A participant was considered to have demonstrated relapse-free efficacy if: a) Participant is slide positive for Plasmodium vivax (P. vivax) at Baseline. b) Participant showed initial clearance of P. vivax parasitemia defined as a negative slide at or before the Day 29 visit. c) Participant is not slide-positive for P. vivax at any assessment. d) Participant did not take a concomitant medication with anti-malarial activity at any point between Study Day 1 and their last parasite assessment. e) Participant is parasite-free at 4 months defined as a negative asexual P. vivax parasite slide at the first parasite assessment performed during study. Microbiologic-Intent-To-Treat (mITT) Population consisted of all participants who received a dose of study treatment (tafenoquine) and had microscopically-confirmed vivax parasitemia at Baseline.
Time Frame: 4 months
Population: mITT Population. Data is not presented for the cohort Tafenoquine 50 mg; as no participants were enrolled in this cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
Number analyzed (Participants) | 14 | 5 | 22 | 19
Participants | 12 | 4 | 20 | 17

8. Secondary Outcome: AUC(0-infinity) of Tafenoquine by Weight Band in Participants Aged >=6 Months to <2 Years (Weighing >=5 kg)
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tafenoquine.
Time Frame: Days 3, 15, 29 and 60 post dose
Population: PK Population. Data is not presented for the cohort Tafenoquine 50 mg; as no participants were enrolled in this cohort.
Arm/Group | Tafenoquine 50 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to Day 120
Description: Safety Population consisted of all participants who received at least one dose of study medication (tafenoquine). All-Cause Mortality, Non-SAEs and SAEs were not collected for tafenoquine 50 mg cohort as no participants were enrolled, because the study sites were unable to find any participants who met the inclusion/exclusion criteria for this cohort.
Groups:
- Tafenoquine 50 mg: Participants with weight band of >=5 to <=10 kg were planned to receive 50 mg tafenoquine on Day 1. Participants were planned to receive Chloroquine according to local/national guidelines to treat the blood stage of Plasmodium vivax.
Arm/Group | Tafenoquine 50 mg | Tafenoquine 100 mg | Tafenoquine 150 mg | Tafenoquine 200 mg | Tafenoquine 300 mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/14 | 0/5 | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/14 | 0/5 | 0/22 | 1/19
Other Adverse Events (participants affected / at risk) | 0/0 | 10/14 | 4/5 | 10/22 | 13/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafenoquine 50 mg (N=0) | Tafenoquine 100 mg (N=14) | Tafenoquine 150 mg (N=5) | Tafenoquine 200 mg (N=22) | Tafenoquine 300 mg (N=19)
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tafenoquine 50 mg (N=0) | Tafenoquine 100 mg (N=14) | Tafenoquine 150 mg (N=5) | Tafenoquine 200 mg (N=22) | Tafenoquine 300 mg (N=19)
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 6
Pyrexia (General disorders) | 0 | 2 | 0 | 5 | 1
Blood methaemoglobin present (Investigations) | 0 | 1 | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT02563496/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT02563496/SAP_001.pdf